CLINICAL TRIAL: NCT04364061
Title: Comparison of Acute Cycling Modalities on Enjoyment, Post Exercise Substrate Oxidation, Appetite and Energy Intakes Over 24h in Postmenopausal Women With Overweight or Obesity
Brief Title: Post Exercise Substrate Oxidation, Appetite and Energy Intakes in Overweight/Obese Postmenopausal Women (EScAPE)
Acronym: EScAPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratoire des Adaptations Métaboliques à l'Exercice en conditions Physiologiques et Pathologiques (Other)
Collaborators: CREPS Auvergne Rhône-Alpes / Vichy (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: IRB00012476-2020-24-03-50
Record Dates: First submitted 2020-04-21; First posted 2020-04-27 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Overweight; Postmenopausal
Keywords: Exercise Modalities; Postmenopausal women; High-intensity interval exercise; CHO and FAT oxidation; Appetite; Energy intakes; Enjoyment
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Masking Description: Data collected on the volunteers will be made anonymous
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Women with overweight or obesity (Experimental)
  Interventions: Other: Moderate Intensity Continuous Exercise; Other: High-Intensity Interval Exercise (1); Other: High-Intensity Interval Exercise (2)

INTERVENTIONS:
Other: Moderate Intensity Continuous Exercise — Participant completed a moderate intensity continuous cycling exercise (MICE) during 35 min at 60-65% thPHRmax
Other: High-Intensity Interval Exercise (1) — Participant completed a high-intensity interval cycling exercise (HIIE 1) during 20min with 60 cycles of speeding up for 8s and pedaling slowly for 12s at 80-90% thPHRmax
Other: High-Intensity Interval Exercise (2) — Participant completed a high-intensity interval cycling exercise (HIIE 2) during 20min with 10 x 1-min bouts at 80-90% thPHRmax, separated by 1-min recovery bouts

SUMMARY:
High-intensity interval exercise (HIIT), as compared to moderate intensity continuous training (MICT), is a time-efficient strategy to decrease total and abdominal fat mass (FM). However, the mechanisms underlying such adaptations are not yet elucidated and research are still needed to establish the optimal HIIT according to subject characteristics. The aim of this study was to compare acute HIIE and MICE cycling exercises on enjoyment, post-exercise substrate oxidation, appetite and energy intakes over 24h in postmenopausal women with overweight or obesity. It is hypothesized that compared with the traditional MICE, HIIE could favor greater enjoyment, higher 2h-post-exercise fat oxidation and a similar energy intakes over 24h despite different post-exercise appetite perceptions.

DETAILED DESCRIPTION:
The aim of this study was to compare acute HIIE and MICE cycling exercises on enjoyment, post-exercise substrate oxidation, and appetite and energy intakes over 24h in postmenopausal women with overweight or obesity.

Using a randomized crossover design, 12 postmenopausal women completed 3 cycling exercises at 6-days intervals:

i) Moderate Intensity Continuous Exercise (MICE) which consisted of 35 min cycling at 60-65% theorical Peak Heart Rate (thPHR) ii) High Intensity Interval Exercise 1 (HIIE 1) 60 cycles of speeding up for 8 s at 80-90%thPHR followed by pedaling slowly for 12 s (20min) iii) High Intensity Interval Exercise 2 (HIIE 2) which consisted of repeated 10 x 1min at 80-90% thPHR followed by pedaling slowly for 1min.

Substrate oxidation (CHO and FAT) were measured at rest and 2h- post exercise. Enjoyment, perceived exertion and appetite were recorded and post-exercise energy intakes were assessed over 24h.

ELIGIBILITY:
Inclusion Criteria:

* postmenopausal women (spontaneous amenorrhea for at least 12 months)
* with overweight or obesity (BMI > 25 kg/m2 and ≤ 40 kg/m2)

Exclusion Criteria:

* medical contraindications to intense physical activity,
* painful joints,
* taking hormone replacement therapy,
* taking B-blockers.

Ages: 50 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Post-exercise (2 hours) CHO and FAT oxidation | 2 hours post-exercise
  CHO and FAT oxidation were measured after each modality with indirect calorimetry during 2 hours post-exercise

SECONDARY OUTCOMES:
Enjoyment | Immediately post-exercise
  Perceive enjoyment evaluated with Physical Activity Enjoyment Scale (PAES) for each modalities. The total scores of PAES are between 18 and 126 with the higher scores indicating greater enjoyment.
Rate Perceive Exertion (RPE) | During exercise (5-10-15 and 20 minutes for HIIE1 and 2 ; 9-18-27 and 35 minutes for MICE) which corresponds at 25-50-75 and 100% of bout completion.
  RPE evaluated with adapted Borg's Scale during exercise for each modalities
Appetite | Before, immediately post-exercise, 60 minutes and 120 minutes post-exercise
  The validated 100 millimeters Visual Analogue Scale (VAS) was used to assess the subjective appetite at 4 time points: before, immediately post-exercise, 60 minutes and 120 minutes post-exercise. This scale comprised four questions anchored with words representing the opposing extreme states of desire to eat, hunger, fullness and prospective food consumption. The score of each question are between 0 and 100.
Energy intakes | 24 hours post-exercise
  Estimated energy intakes using dietary questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Claire MOREL, Dr, Principal Investigator — CREPS Auvergne Rhône-Alpes / Vichy
Locations (1):
- CREPS Auvergne Rhône-Alpes / Vichy, Bellerive-sur-Allier, Allier, France